CLINICAL TRIAL: NCT04070599
Title: Predictive Value of the Initial Hemato-immunological Profile on the Evolution of Immunological Thrombopenic Purpura of Children and Adults.
Brief Title: Initial Hemato-immunological Profile on the Evolution of Immunological Thrombopenic Purpura.
Acronym: IMMUNOTI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2010/30
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Immune Thrombocytopenic Purpura; Autoimmune Thrombocytopenia; Thrombopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Study of lymphocyte subpopulations, cytokine assays, identification of autoantibodies, study of CD40 platelet ligand, thrombopoietin assay
  Interventions: Biological: Collection of biological samples

INTERVENTIONS:
Biological: Collection of biological samples — A collection of biological samples will be carried out, with the remainders of the immunological samples taken on dry tube: the serum of the patients, taken at the initial diagnosis, will be kept frozen at -20 ° C.

SUMMARY:
This study aims to determine the hemato-immunological parameters predictive of the evolution of a Immune thrombocytopenic purpura (ITP) towards chronicity, and to identify possible differences between the child and the adult.

DETAILED DESCRIPTION:
Immune thrombocytopenic purpura (ITP) is a rare autoimmune thrombocytopenia whose incidence is 2 to 5 cases / 100,000 inhabitants / year. The potentially serious haemorrhagic risk is the major issue of management. A recent international consensus conference classifies PTI according to the duration of thrombocytopenia: acute ITP (<3 months), persistent ITP (3-12 months) and chronic ITP (> 12 months) (Rodeghiero 2009). In the acute or persistent phase, polyvalent immunoglobulins (IVIG) and / or corticosteroids are proposed. In the chronic phase, splenectomy is a possible cure for 70% of patients. No predictor of treatment response is known.

The pathophysiology of ITP is multifactorial: platelet phagocytosis, mediated by autoantibody, macrophages of the reticuloendothelial system, and destruction in the spleen, genetic background and / or environmental factor favoring the role of certain lymphocyte subpopulations, cytotoxic or regulatory T, via their cytokine environment, abnormalities of thrombopoiesis.

ITP affects children as well as adults, but the evolutionary profile is very different. In children, ITP, which is often post-infectious, is acute in 80% of cases, whereas ITP in adults has a chronic evolution in 80% of cases. The primary diagnostic and therapeutic practices are similar. The reasons for these evolutionary differences are not known and little studied.

Is the orientation of the hemato-immunological response observed during the first episode of ITP different in children and adults? Do these differences explain the evolutionary specificities of the two age groups? Are there hematologic parameters predictive of a response to initial treatments?

ELIGIBILITY:
Inclusion Criteria:

* Minor patients aged 2 to 18 recruited at the Children's Hospital, in the service of Prof. Y. PEREL, Dr. N. ALADJIDI, CEREVANCE,
* Adult patients (> 18 years old) recruited at the Haut-Lévêque hospital, Pr JL PELLEGRIN, Pr JF VIALLARD, GECAI,
* Patient with acute Immune thrombocytopenic purpura, seen at initial diagnosis or within 8 days (defined as thrombocytopenia <100 G / L, after an infectious cause, drug or related to autoimmune disease, hematological malignancy or deficit Immune have been eliminated, Rodeghiero criteria, 2009).
* Patient who received immunoglobulins more than 4 weeks before inclusion
* Written consent given by the patient, if he is of age, or by the person (s) having parental authority
* Patient affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Patient who has received specific treatment from an Immune thrombocytopenic purpura
* Patient with secondary Immune thrombocytopenic purpura (hematological malignancy, autoimmune disease, immunodeficiency, pregnancy)
* Patient placed under the protection of justice

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-04-12 (Actual); Primary Completion 2014-03-05 (Actual); Study Completion 2014-03-05 (Actual)

PRIMARY OUTCOMES:
Complete remission yes/no | At 12 months of initial diagnosis
  The status of Immune thrombocytopenic purpura in adult and pediatric patients will be determined at 12 months of initial diagnosis according to the Rodeghiero criteria: complete remission if the platelet count is> 100 G / L. A non-complete remission patient at 12 months will be considered to have a chronic Immune thrombocytopenic purpura.

SECONDARY OUTCOMES:
Response to the first course of first-line treatments (Immunoglobulin IV or corticosteroid) | At Day14
  Defined by the Rodeghiero criteria: complete response (platelet count> 100 G / L and no bleeding), response (platelet count> 30 G / L and increase> 2 times the basal rate and no bleeding), no response (platelet count <30 G / L or increase <2 times the basal rate or bleeding).
Response to the first course of first-line treatments (Immunoglobulin IV or corticosteroid) | At Day 28
  Defined by the Rodeghiero criteria: complete response (platelet count> 100 G / L and no bleeding), response (platelet count> 30 G / L and increase> 2 times the basal rate and no bleeding), no response (platelet count <30 G / L or increase <2 times the basal rate or bleeding).

CONTACTS AND LOCATIONS:
Overall Officials: Carine GRIEB, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No